CLINICAL TRIAL: NCT00832819
Title: E7080 in Combination With Carboplatin and Paclitaxel in Patients With Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-J081-110
Record Dates: First submitted 2009-01-23; First posted 2009-01-30 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-02

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Cancer; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms | interventions — lenvatinib; Paclitaxel; Carboplatin

ARMS (2):
- E7080 (Dose Escalation Cohort) (Experimental): This will be a dose-escalation evaluation of 12-18 participants to determine the maximum tolerated dose of E7080 in combination with paclitaxel and carboplatin.
  Interventions: Drug: E7080; Drug: Paclitaxel; Drug: Carboplatin
- E7080 (Expansion Cohort) (Experimental): Dosage of E7080 for Expansion Cohort will be determined based on the maximum tolerated dose in the Dose-Escalation Cohort.
  Interventions: Drug: E7080; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: E7080 — Drug: E7080 will be administered orally starting at a dose of 6 mg twice daily during the 7-day run-in period and for 3 weeks (Cycle 1).
  Arms: E7080 (Dose Escalation Cohort)
Drug: E7080 — Maximum tolerated dose determined in the Dose-Escalation Cohort will be administered to the Expansion Cohort. After E7080 is taken on Day 1, paclitaxel (200 mg/m2) will be administered intravenously (IV), followed by IV carboplatin (AUC 6.0 min/mg/mL).
  Arms: E7080 (Expansion Cohort)
Drug: Paclitaxel — Paclitaxel (200 mg/m2) will be administered intravenously (IV) on Day 1 after administration of E7080.
Drug: Carboplatin — Carboplatin (AUC 6.0 min/mg/mL) will be administered IV on Day 1 after administration of E7080 and Paclitaxel.

SUMMARY:
The purpose of this study is to determined the maximum tolerated dose (MTD), safety and tolerability, pharmacokinetics, pharmacodynamics, and anti-tumor effect of E7080 administered continually twice daily in combination with carboplatin and paclitaxel to patients with advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion criteria:

1. Subjects with a histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC).
2. Locally advanced and/or metastatic non-small cell lung cancer (NSCLC) (Stage IIIB/IV).
3. Subjects with at least one measurable tumor lesion by Response Evaluation Criteria In Solid Tumors (RECIST).
4. Subjects with Performance Status (PS) 0-1.
5. Subjects with adequate organ function.

Exclusion criteria:

1. Subjects who have ever received the following therapy for non-small cell lung cancer (NSCLC):

   1. Chemotherapy
   2. Biological or immunotherapies
   3. Surgery for primary focus
   4. The radiation therapy for primary focus
2. Subjects with the severe complications or disease history.
3. Subjects with brain metastasis accompanying clinical symptoms or requiring treatment.
4. Subjects with simultaneous or metachronous cancers.
5. Subjects who cannot take oral medication.
6. Subjects who are using drugs that strongly inhibit or induce cytochrome P450 (CYP) 3A4.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wataru Yusa, Study Director — Oncology Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (3):
- Japan (3):
  - Sunto-gun, Shizuoka
  - Chuo-ku, Tokyo
  - Koto-ku, Tokyo

REFERENCES:
- [Derived] Nishio M, Horai T, Horiike A, Nokihara H, Yamamoto N, Takahashi T, Murakami H, Yamamoto N, Koizumi F, Nishio K, Yusa W, Koyama N, Tamura T. Phase 1 study of lenvatinib combined with carboplatin and paclitaxel in patients with non-small-cell lung cancer. Br J Cancer. 2013 Aug 6;109(3):538-44. doi: 10.1038/bjc.2013.374. Epub 2013 Jul 16. PMID 23860537

RESULTS

PARTICIPANT FLOW:
Groups:
- E7080 4 mg BID (Dose Escalation): E7080 mono-therapy (initial dose was 4 mg BID) was orally administered twice daily for 7 days in run-in period (Cycle 0); subsequently from Cycle 1 but up to 6 Cycles, E7080 treatment was continued with the combination of carboplatin (AUC 6.0 min/mg/mL) and paclitaxel (200 mg/m2) on Day 1 every 3 weeks.
- E7080 6 mg BID (Dose Escalation): E7080 mono-therapy (initial dose was 6 mg BID) was orally administered twice daily for 7 days in run-in period (Cycle 0); subsequently from Cycle 1 but up to 6 Cycles, E7080 treatment was continued with the combination of carboplatin (AUC 6.0 min/mg/mL) and paclitaxel (200 mg/m2) on Day 1 every 3 weeks.
- E7080 4 mg BID (Expansion): Dosage of E7080 for expansion cohort was determined based on the maximum tolerated dose (MTD). The MTD for E7080 with with the combination of carboplatin and paclitaxel was 4 mg BID (Arm 1). For the expansion cohort, run-in treatment (Cycle 0) was not performed and E7080 treatment (4 mg BID) began from Cycle 1 but up to 6 Cycles with the combination of carboplatin (AUC 6.0 min/mg/mL) and paclitaxel (200 mg/m2) on Day 1 every 3 weeks.
Period: Overall Study
Arm/Group | E7080 4 mg BID (Dose Escalation) | E7080 6 mg BID (Dose Escalation) | E7080 4 mg BID (Expansion)
Started | 6 | 6 | 16
Completed | 6 | 5 | 15
Not Completed | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- E7080 4 mg BID (Dose Escalation): E7080 mono-therapy (initial dose was 4 mg BID) was orally administered twice daily for 7 days in run-in period (Cycle 0); subsequently from Cycle 1 but up to 6 Cycles, E7080 treatment was continued with the combination of carboplatin (Area under the curve (AUC) 6.0 min/mg/mL) and paclitaxel (200 mg/m2) on Day 1 every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | E7080 4 mg BID (Dose Escalation) | E7080 6 mg BID (Dose Escalation) | E7080 4 mg BID (Expansion) | Total
Number analyzed (Participants) | 6 | 6 | 16 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (9.3) | 54.8 (9.7) | 58.4 (11.2) | 56.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 4 | 4 | 13 | 21

OUTCOME MEASURES:

1. Secondary Outcome: Anti-tumor Effect of E7080 in Combination With Carboplatin and Paclitaxel.
Time Frame: At Screening, on Day 22 of every even cycle, and at discontinuation
Reporting Status: Not Posted

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Tolerability was confirmed by the frequency of occurrence of Dose Limiting Toxicities (DLTs) observed by the end of Cycle 1 in 6 participants.
Time Frame: 7 days during the run-in period (Cycle 0) and 3 weeks (21 days) from Cycle 1
Population: DLTs were analyzed on the Safety Analysis Set; however subjects with 75% or less treatment compliance for E7080 in Cycle 1 or those who discontinued the study and had no confirmed data on tolerability up to Cycle 1 Day 22 were excluded from this analysis.
Measure: Number; unit: mg BID
Arm/Group | E7080 6 mg BID (Dose Escalation)
Number analyzed (Participants) | 6
mg BID | 4

3. Secondary Outcome: Pharmacokinetics and Pharmacodynamics of E7080 in Combination With Carboplatin and Paclitaxel.
Time Frame: At various time points until Day 22 of Cycle 1
Reporting Status: Not Posted

4. Secondary Outcome: To Evaluate the Safety and Tolerability of E7080 in Combination With Carboplatin and Paclitaxel.
Description: Refer safety section for safety analysis
Time Frame: Throughout the study until 30 days after last dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout the study until 30 days after last dose
Description: All participants who received at least one E7080 dose and had evaluable data were included in the safety analyses.
Arm/Group | E7080 4 mg BID (Dose Escalation) | E7080 6 mg BID (Dose Escalation) | E7080 4 mg BID (Expansion)
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 6/16
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7080 4 mg BID (Dose Escalation) (N=6) | E7080 6 mg BID (Dose Escalation) (N=6) | E7080 4 mg BID (Expansion) (N=16)
Syncope (Nervous system disorders) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Metastatses to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7080 4 mg BID (Dose Escalation) (N=6) | E7080 6 mg BID (Dose Escalation) (N=6) | E7080 4 mg BID (Expansion) (N=16)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 13
Erythropenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 6 | 5 | 15
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 10
Neutropenia (Blood and lymphatic system disorders) | 6 | 5 | 15
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4 | 16
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 2 | 4 | 7
Thyroiditis subacute (Endocrine disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Anal erosion (Gastrointestinal disorders) | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 4 | 12
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 12
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 2
Gingival discolouration (Gastrointestinal disorders) | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 2 | 0 | 4
Nausea (Gastrointestinal disorders) | 5 | 6 | 13
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 1 | 2
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 2 | 7
Vomiting (Gastrointestinal disorders) | 2 | 3 | 8
Chest pain (General disorders) | 0 | 1 | 0
Extravasation (General disorders) | 0 | 0 | 2
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 5 | 5 | 10
Impaired healing (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 3 | 7
Anal abscess (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3
Oral herpes (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 3
Pneumonia (Infections and infestations) | 1 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 3 | 8
Aspartate aminotransferase increased (Investigations) | 4 | 6 | 5
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 3
Blood creatinine increased (Investigations) | 1 | 1 | 4
Blood lactate dehydrogenase increased (Investigations) | 2 | 1 | 4
Blood thyroid stimulating hormone increased (Investigations) | 3 | 0 | 5
Blood urea increased (Investigations) | 2 | 0 | 5
Blood urine present (Investigations) | 2 | 3 | 5
C-reactive protein increased (Investigations) | 2 | 0 | 3
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 2 | 5
Haemoglobin decreased (Investigations) | 2 | 0 | 2
Occult blood (Investigations) | 0 | 0 | 1
Protein total decreased (Investigations) | 1 | 1 | 5
Weight decreased (Investigations) | 3 | 5 | 8
Weight increased (Investigations) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4 | 13
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 3 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 3 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 11
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 8
Head discomfort (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 8
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 5 | 15
Depression (Psychiatric disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 4
Glycosuria (Renal and urinary disorders) | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 6 | 3 | 11
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Penile haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 5 | 15
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 5 | 12
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Angiopathy (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 2 | 1 | 2
Hypertension (Vascular disorders) | 5 | 5 | 11
Hypotension (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other